CLINICAL TRIAL: NCT01497873
Title: A Phase IIb, Randomized, Open, Parallel-Group, Multi-Center Trial to Assess the Efficacy and Safety of Belotecan(CamtoBell Inj.) or Topotecan in Patients With Relapsed Small Cell Lung Cancer
Brief Title: A Randomized Study to Compare the Efficacy and Safety of Belotecan and Topotecan as Monotherapy for Sensitive-Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11SCLC09I
Record Dates: First submitted 2011-04-20; First posted 2011-12-23 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; Belotecan; Topotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; belotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Belotecan (Experimental): Camtobell Injection
  Interventions: Drug: Belotecan
- Topotecan (Active Comparator): Hycamtin Injection
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Topotecan — 1.5 mg/m^2 IV days 1, 2, 3, 4, 5 of each 21-day cycle until 6 cycle or more
  Other Names: Hycamtin Injection
  Arms: Topotecan
Drug: Belotecan — 0.5 mg/m^2 IV days 1, 2, 3, 4, 5 of each 21-day cycle until 6 cycle or more
  Other Names: Camtobell Injection
  Arms: Belotecan

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Belotecan administered 5 days every 3 weeks in comparison to Topotecan in Patients with relapsed small cell lung cancer.

DETAILED DESCRIPTION:
A Phase Ⅱb, Randomized, Open, Parallel-Group, Multi-Center Trial to Assess the Efficacy and Safety of Belotecan(CamtoBell inj.) or Topotecan in Patients with Relapsed Small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histological or cytological diagnosis of SCLC
* Limited disease (LD) or Extensive disease (ED) at time of study entry
* Recurrent or progressive SCLC ≥ 90 days of duration of response for firstline therapy
* Measurable disease defined by RECIST criteria
* ECOG Performance Status of 0, 1, or 2
* Life expectancy ≥ 3 months
* Adequate bone marrow, Renal, Hepatic reserve:

absolute neutrophil (segmented and bands) count (ANC) ≥ 1500 cells/mm3 platelet count ≥ 100,000 cells/ mm3 hemoglobin ≥ 9 g/dL Total bilirubin ≤ 1.5 mm3 Alanine aminotransferase (ALT) and aspartate aminotransferase(AST) ≤ 2.0 X ULN Alkaline Phosphatase (ALP) ≤ 2.0 X ULN Serum creatinine ≤ 1.5mg/dL or calculated creatinine clearance > 60mL/min

- Signed a written informed consent

Exclusion Criteria:

* Active infection
* Symptomatic brain lesion
* Any other type of cancer during the previous 5 years
* Severe concurrent diseases
* Prior anticancer therapy within 4 weeks before enroll
* Active pregnancy test and Pregnant or nursing women
* Participation in any investigational drug study within 28 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Objectives Response Rate(ORR, %) | Up to 18weeks
  The response rate was defined as the test subject who had a complete response (CR) or a partial response (PR) as determined by the 'tumor response evaluation' criteria specified in the research protocol

SECONDARY OUTCOMES:
Overall Survival(OS) | 7years
  Defined as the time from the randomization to the time of death.
Progression Free survival(PFS) | Up to 18weeks
  Defined as the elapsed time from the time of randomization to the time of confirmation of progression or the time of death

CONTACTS AND LOCATIONS:
Overall Officials: Heung Tae Kim, M.D., Ph.D, Principal Investigator — National Cancer Center; Jin Hyoung Kang, M.D., Ph.D, Principal Investigator — The Catholic University of Korea Seoul St. Marys Hospital; Jin Young Kim, M.D., Ph.D, Principal Investigator — Keimyung University Dongsan Medical Center; Dong-Wan Kim, M.D., Ph.D, Principal Investigator — Seoul National University Hospital; Sang-We Kim, M.D., Ph.D, Principal Investigator — Asan Medical Center; Hye Ryeon Kim, M.D., Ph.D, Principal Investigator — Yonsei Cancer Center; Jin Hyuk Choi, M.D., Ph.D, Principal Investigator — Ajou University School of Medicine; Ki Hyeong Lee, M.D., Ph.D, Principal Investigator — Chungbuk National University Hospital; Ho Jung An, M.D., Ph.D, Principal Investigator — St. Vincents Hospital; Chi Hoon Maeng, M.D., Ph.D, Principal Investigator — Kyung Hee University Medical Hospital; Jin-Soo Kim, M.D., Ph.D, Principal Investigator — SMG-SNU Boramae Medical Center; Joung Soon Jang, M.D., Ph.D, Principal Investigator — Choung Ang University Hospital; Bong Seog Kim, M.D., Ph.D, Principal Investigator — Seoul Veterans Hospital; Joo-Hang Kim, .D., Ph.D, Principal Investigator — CHA Bundang Medical Center
Locations (14):
- South Korea (14):
  - Chungbuk University Hospital, Daegu
  - Keimyung University Dongsan Center, Daegu
  - National Cancer Center, Goyang
  - Asan Medical Center, Seoul
  - CHA Bundang Medical Center, Seoul
  - Chung-Ang University hospital, Seoul
  - Kyung Hee University Medical Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Marys Hospital, Seoul
  - Seoul Veterans Hospital, Seoul
  - Yonsei Cancer Center, Seoul
  - Ajou University Hospital, Suwon
  - St. Vincents Hospital, Suwon

REFERENCES:
- [Derived] Kang JH, Lee KH, Kim DW, Kim SW, Kim HR, Kim JH, Choi JH, An HJ, Kim JS, Jang JS, Kim BS, Kim HT. A randomised phase 2b study comparing the efficacy and safety of belotecan vs. topotecan as monotherapy for sensitive-relapsed small-cell lung cancer. Br J Cancer. 2021 Feb;124(4):713-720. doi: 10.1038/s41416-020-01055-5. Epub 2020 Nov 16. PMID 33191408